CLINICAL TRIAL: NCT05723952
Title: Effect of Barcelona Scoliosis Physical Therapy Versus International Scoliosis Schroth Therapy in Adolescent Idiopathic Scoliosis
Brief Title: Effect of Barcelona School and Schroth for Adolescent Idiopathic Scoliosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Mahmoud sherf eldin, master student, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EG,KFS lab research
Record Dates: First submitted 2022-12-23; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Idiopathic Scoliosis, Thoracic Region

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barcelona scoliosis physical therapy school (Experimental): procedure for treating scoliosis
  Interventions: Other: Barcelona scoliosis physical therapy school
- International scoliosis schroth therapy (Experimental): procedure for treating scoliosis
  Interventions: Other: International scoliosis schroth therapy

INTERVENTIONS:
Other: Barcelona scoliosis physical therapy school — procedure for treating Adolescent Idiopathic scoliosis
  Arms: Barcelona scoliosis physical therapy school
Other: International scoliosis schroth therapy — procedure for treating Adolescent Idiopathic scoliosis
  Arms: International scoliosis schroth therapy

SUMMARY:
for adolescent idiopathic scoliosis child, investigator will use Barcelona scoliosis physical therapy school and International scoliosis schroth therapy to see which school is better in dealing with scoliosis.

ELIGIBILITY:
Inclusion Criteria:

scoliosis with angle < 25 participant has Risser sign of П-V participant is not receiving other treatment during study participant not using braces or muscle relaxants

Exclusion Criteria:

scoliosis due to congenital, neuro-muscular, or syndromic etiology, participant who has true leg length discrepancy participant who has cardiac anomalies participant who has kyphosis.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Cobb's Angle | 3 month
  to determine angle of scoliosis
Angle Trunk Rotation (ATR): | 3 month
  to determine amount of hump

SECONDARY OUTCOMES:
SRS-22 patient questionnaire | 3 month
  questionnaire to evaluate pain for spinal deformity patient

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
share the result of the study not any personal information about patient